CLINICAL TRIAL: NCT02135770
Title: Randomized Control Trial to Assessed the Impact of Low Dose Unfractionated Heparin Treatment on Inflammation in Severe Sepsis
Brief Title: Impact of Low Dose Unfractionated Heparin Treatment on Inflammation in Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Khie Chen Lie, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLDS01
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Severe Sepsis With Septic Shock; Severe Sepsis Without Septic Shock
Keywords: heparin; sepsis; inflammation
MeSH Terms: conditions — Sepsis; Inflammation | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unfractionated Heparin (Experimental): Low dose unfractionated Heparin 10 unit/kgBW/hour continuous infusion
  Interventions: Drug: Unfractionated heparin
- Placebo (Placebo Comparator): Normal saline packed in same form with trial drugs.

INTERVENTIONS:
Drug: Unfractionated heparin — 10 unit/kgBW/hour continuous infusion for 72 hours
  Arms: Unfractionated Heparin

SUMMARY:
Sepsis is a clinical syndrome which infection trigger systemic inflammatory response. Uncontrolled inflammatory process leads to multiple organ dysfunction and cause early mortality in severe sepsis. Unfractionated heparin is an anticoagulant that widely used either for DVT prophylaxis or treatment of disseminated intravascular coagulation. Heparin also have an anti-inflammatory effect through downregulates nuclear factor kappa B and tumor necrosis factor alpha.

Aim of this study is to determine effects of low dose unfractionated heparin treatment on inflammation in severe sepsis patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe sepsis and septic shock define by revised Sepsis Criteria (2001)
* Within 48 hour diagnose sepsis
* Agree to participate

Exclusion Criteria:

* Pregnancy and lactation
* Severe thrombocytopenia, platelet less than 30.000/mm3
* Bleeding or high risk of major bleeding
* During anticoagulant treatment
* After thrombolytic treatment
* Decompensated chronic liver diseases
* Chronic kidney diseases on dialysis treatment
* During high dose corticosteroid treatment
* HIV with CD4 count below 50/mm3
* Indication for high dose heparin treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
inflammation | 3 days
  determine effects of low dose unfractionated heparin treatment on nuclear factor kappa B, inhibitor kappa B kinase and tumor necrosis factor-alpha.

SECONDARY OUTCOMES:
clinical outcome | 14 days
  determine impact of low dose unfractionated heparin on mortality and improvement APACHE II score

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Cipto Mangunkusumo General Hospital, Jakarta, Indonesia